CLINICAL TRIAL: NCT04796480
Title: Comparison Of Outcome Of Lactose Free Formula Milk With Yogurt In Children With Acute Diarrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Services Hospital, Lahore (Other Government)
Responsible Party: Principal Investigator, Dr. Mahjabeen Akram, Principal Investigator, Services Hospital, Lahore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HOSPITAL
Record Dates: First submitted 2021-03-08; First posted 2021-03-15 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Acute Diarrhea
Keywords: LACTOSE FREE FORMULA MILK; YOGURT
MeSH Terms: interventions — Yogurt

STUDY DESIGN:
Intervention Model Description: Participants were divided in 2 groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- YOGURT (Active Comparator): Group 1 children were given home made plain yogurt in treatment of acute diarrhea
  Interventions: Dietary Supplement: YOGURT
- LACTOSE FREE FORMULA MILK (Active Comparator): Group 2 children were given lactose free formula milk in treatment of acute diarrhea
  Interventions: Dietary Supplement: LACTOSE FREE FORMULA MILK

INTERVENTIONS:
Dietary Supplement: YOGURT — Group 1 was given yogurt
  Arms: YOGURT
Dietary Supplement: LACTOSE FREE FORMULA MILK — Group 2 was given lactose free formula milk
  Arms: LACTOSE FREE FORMULA MILK

SUMMARY:
This study was aimed to look at the effect of lactose free formula milk in comparison with home-made plain yogurt in children with acute watery diarrhea.

DETAILED DESCRIPTION:
A randomized controlled trial using non probability consecutive sampling was carried out on 60 children (30 in each group) in Department of Paediatrics Unit I, Services Hospital Lahore. An informed written consent was taken from parents of the children. Ethical issues considered and maintained throughout the study. Then all children were randomly divided in two groups by using lottery method. In group 1; children were given yogurt while in group 2, children were given lactose free formula milk. In both groups, feed was given 5-8 times per day. Patients were followed-up till resolution of symptoms and discharge from hospital.

ELIGIBILITY:
Inclusion Criteria:

* Children of age 4-24 months presenting with acute diarrhea
* Both gender

Exclusion Criteria:

* Children on antibiotic therapy within 48 hours prior to presentation
* Malnourished children (-2SD as per WHO criteria)
* Children with severe dehydration requiring IV fluids
* Children < 4 months of age (as weaning not started yet)

Ages: 4 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2018-06-10 (Actual); Primary Completion 2018-12-09 (Actual); Study Completion 2018-12-09 (Actual)

PRIMARY OUTCOMES:
Effect of home-made yogurt versus lactose-free milk on mean duration of diarrhea in children with acute diarrhea | 6 Months
  The effect of home-made yogurt and lactose-free milk in children with acute diarrhea was compared i.e. to check out which one is more suitable to treat diarrhea by measuring the mean duration of diarrhea in hours. The reason behind the effectiveness of yogurt against lactose-free milk is the presence of probiotics within it, which help in recovering of good bacteria population in intestine and so may help in decreasing duration and severity of diarrhea.

CONTACTS AND LOCATIONS:
Locations (1):
- Services Hospital Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kosek M, Bern C, Guerrant RL. The global burden of diarrhoeal disease, as estimated from studies published between 1992 and 2000. Bull World Health Organ. 2003;81(3):197-204. Epub 2003 May 16. PMID 12764516
- [Background] Chu C, Rotondo-Trivette S, Michail S. Chronic diarrhea. Curr Probl Pediatr Adolesc Health Care. 2020 Aug;50(8):100841. doi: 10.1016/j.cppeds.2020.100841. Epub 2020 Aug 27. PMID 32863166
- [Background] Forster CS, Hsieh MH, Cabana MD. Perspectives from the Society for Pediatric Research: Probiotic use in urinary tract infections, atopic dermatitis, and antibiotic-associated diarrhea: an overview. Pediatr Res. 2021 Aug;90(2):315-327. doi: 10.1038/s41390-020-01298-1. Epub 2020 Dec 7. PMID 33288875